CLINICAL TRIAL: NCT04646902
Title: Relevance of the Ratio Kynurenine/Tryptophan to Characterize Hypertension Associated to Obstructive Sleep Apnea (KYNTOSA)
Brief Title: Kynurenine/Tryptophan Ratio in Hypertension Associated to Obstructive Sleep Apnea
Acronym: KYNTOSA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Universidade Nova de Lisboa (Other)
Collaborators: Centro Hospitalar Lisboa Ocidental (Other Government); Centro Hospitalar de Lisboa Central (Other); Hospital Beatriz Ângelo (Other); Hospital Fernando Fonseca (Unknown); Hospital da Luz, Portugal (Other)
Responsible Party: Sponsor
Other Study IDs: Kyntosa_02_20200428; PTDC/MED-TOX30418/2017 (Other Grant/Funding Number: Fundação para a Ciência e a Tecnologia)
Record Dates: First submitted 2020-10-12; First posted 2020-11-30 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Hypertension Secondary
Keywords: hypertension; obstructive sleep apnea; tryptophan; aryl hydrocarbon receptor
MeSH Terms: conditions — Hypertension; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Serum samples Urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- HTN_OSA: Patients with hypertension* with obstructive sleep apnea**
  * Hypertension will be defined as: i) use of antihypertensive drug(s) and stable dose for at least 2 weeks prior to inclusion; or ii) in untreated patients: office systolic blood pressure values >= 140 mmHg and/ or diastolic blood pressure values >= 90 mmHg.
  ** OSA will be defined with a polysomnography level 1, 2 or 3 performed within the previous twelve months with:
  * an apnea-hypopnea index > 5 events per hour (with more than 50% of obstructive events) associated with symptoms (associated sleepiness, fatigue, insomnia, snoring, subjective nocturnal respiratory disturbance or observed apnea) or medical/psychiatric disorder (hypertension, coronary artery disease, atrial fibrillation, congestive heart failure, stroke, diabetes, cognitive dysfunction, or mood disorder), OR
  * an apnea-hypopnea index > 15 events per hour, AND
  * no significant changes in health, medications, or lifestyle since the polysomnography.
- HTN_NoOSA: Patients with hypertension without obstructive sleep apnea
- NoHTN_OSA: Patients without hypertension with obstructive sleep apnea
- NoHTN_NoOSA: Patients without hypertension without obstructive sleep apnea (healthy controls)

SUMMARY:
Obstructive Sleep Apnea (OSA) is an independent risk factor for hypertension (HTN) and the most common cause of resistant HTN. The mechanisms underlying OSA-associated HTN are not completely understood. This is crucial to find novel therapeutic targets of OSA-associated HTN. The Aryl Hydrocarbon Receptor (AHR) is a cytosolic transcription factor that has been linked with the pathogenesis of HTN.

This study aims to evaluate the role of endogenous ligands of AHR such as kynurenine in discriminating patients with OSA-associated HTN. For that aim, a case-control study will be performed in patients with and without hypertension exposed and not exposed to OSA. Kynurenine and other metabolites will be quantified in urine and serum samples.

ELIGIBILITY:
CASES (subjects with hypertension with and without OSA)

Inclusion Criteria:

* Adults ≥ 30 years old attending the outpatient clinics of the clinical sites.
* Diagnosis of hypertension defined either as: a) use of antihypertensive drug(s) and stable dose for at least 2 weeks prior to inclusion; or b) in untreated patients: office systolic blood pressure values >= 140 mmHg and/ or diastolic blood pressure values >= 90 mmHg.
* Able to understand and communicate effectively with study personnel.
* Giving written informed consent to participate.

Exclusion Criteria:

* Self-reported pregnancy or breastfeeding.
* Patients on haemodialysis or peritoneal dialysis.
* Chronic liver disease with Child-Pugh score B or higher.
* Hypertension attributed to renal artery stenosis, primary hyperaldosteronism, pheochromocytoma, Cushing's syndrome, coarctation of aorta.
* History of any OSA surgical treatment to the palatal and hypopharyngeal regions, notably uvulopalatopharyngoplasty surgery (UPPP), palatal radio frequency ablation, tonsillectomy, lingual tonsillectomy, partial glossectomy, tongue base radio frequency ablation, genioglossal advancement, hyoid suspension, maxillomandibular advancement surgery (MMA) and active use of hypoglossal nerve stimulator.
* Patients with a good adherence to CPAP, defined as the use of CPAP for at least 4 hours/night on 70% of nights during the last 3 months.
* Pulmonary hypertension.
* Current diagnosed oncological disease.
* Patients with known chronic or acute infectious diseases.
* Other current severe progressive or uncontrolled disease which in the judgement of the investigator renders the patient unsuitable for the study

CONTROLS (individuals without hypertension with and without OSA) For each case, an age and gender-matched control will be selected.

Exclusion Criteria:

* Pregnancy or breastfeeding.
* Patients on haemodialysis or peritoneal dialysis.
* Chronic liver disease with Child-Pugh score b or higher.
* History of any OSA surgical treatment to the palatal and hypopharyngeal regions, notably uvulopalatopharyngoplasty surgery (UPPP), palatal radio frequency ablation, tonsillectomy, lingual tonsillectomy, partial glossectomy, tongue base radio frequency ablation, genioglossal advancement, hyoid suspension, maxillomandibular advancement surgery (MMA) and active use of hypoglossal nerve stimulator.
* Patients with a good adherence to CPAP, defined as the use of CPAP for at least 4 hours/night on 70% of nights during the last 3 months.
* Pulmonary hypertension.
* Current diagnosed oncological disease.
* Patients with known chronic or acute infectious diseases.
* Patients with known chronic or acute infectious diseases.
* Other current severe progressive or uncontrolled disease which in the judgement of the investigator renders the patient unsuitable for the study.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include 4 groups of adults: healthy volunteers; normotensive OSA patients; hypertensive OSA patients; hypertensive non OSA patients.
Sampling Method: Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Kynurenine / Tryptophan ratio | Day 1 (visit 1)
  Ratio between kynurenine and tryptophan concentrations

SECONDARY OUTCOMES:
Concentrations of metabolites | Day 1 (visit 1)
  The relevant metabolites and their concentration will be identified by Partial Least Square Discriminant Analysis (PLS-DA) applied to non-targeted metabolomics.

CONTACTS AND LOCATIONS:
Overall Officials: Maria E Monteiro, PhD, Principal Investigator — Universidade NOVA Lisboa
Locations (5):
- Portugal (5):
  - Centro Hospitalar de Lisboa Central, Lisbon
  - Centro Hospitalar Lisboa Ocidental, Lisbon
  - Hospital Beatriz Ângelo, Lisbon
  - Hospital da Luz, Lisbon
  - Hospital Fernando Fonseca, Lisbon

IPD SHARING:
Plan to Share IPD: No